CLINICAL TRIAL: NCT05700513
Title: The Joint Effects of Dog-rose, Cranberry Leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, and Sumac for Controlling Blood Glucose of Patients With Type II Diabetes Mellitus: A Phase 1-2 Randomized Placebo-Controlled Trial
Brief Title: Dog-rose, Cranberry Leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica and Sumac in Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Principal Investigator, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70746
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Insulin resistance; Lipochromin; Vaccinium macrocarpon; Medicago sativa; Trigonella; Fenugreek; Lemon Beebrush; Urtica dioica; Rhus; Sumac
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsules containing the combination products (Active Comparator): Capsules containing dog-rose, Cranberry leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, and Sumac
  Interventions: Combination Product: Capsules containing the combination products
- Placebo (Placebo Comparator): Placebo capsules containing maltodextrin
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Combination Product: Capsules containing the combination products — Capsules containing dog-rose, Cranberry leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, and Sumac
  Arms: Capsules containing the combination products
Drug: Placebo capsules — Placebo capsules containing maltodextrin
  Arms: Placebo

SUMMARY:
This study investigates the safety and combined effect of Cranberry leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, Dog-rose, and Sumac on improving the glycemic profile of patients with type 2 diabetes mellitus compared to the placebo group.

DETAILED DESCRIPTION:
The present double-blind, randomized and placebo-controlled study will be conducted on type 2 diabetes mellitus patients to evaluate the safety and combined effect of Cranberry leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, Dog-rose, and Sumac on improving glycemic profiles (fasting blood sugar, glycosylated Hemoglobin, 2 hours postprandial blood sugar, insulin concentration, insulin resistance, and beta-cell function). The study also evaluates systolic blood pressure, diastolic blood pressure, anthropometric variables, lipid profile, C-reactive protein, and renal and liver function tests.

A pilot study with 30 participants will be conducted to estimate the sample size considering 0.05 first type error and a power of 80%. Individuals aged between 18-70 with a diagnosis of type 2 diabetes mellitus based on WHO criteria for at least one year will be enrolled. Participants will be randomized in the placebo or intervention group to receive two capsules per day before lunch and dinner for six months containing 200 milligrams of equally combined extracts of Cranberry leaves, Cranberry Berries, Alfalfa, Fenugreek, Lemon Beebrush, Urtica, Dog-rose, and Sumac. Participants will be followed up with four office visits (t0= baseline, 1=15th day, 2t=3rd month, 3t=6th month) to assess outcomes. Also, the complications and adherence of patients to intervention will be checked every two weeks by telephonic discussion. The analysis will be performed based on the intent-to-treat method.

ELIGIBILITY:
Inclusion Criteria:

* At least one year of diagnosis of type 2 diabetes according to the criteria of the World Health Organization,
* Hemoglobin A1c (HbA1c) > 7.0% or fasting blood glucose > 7.0 mmol/L,
* Body mass index (BMI) more than 23 kg/m2 and less than 35.

Exclusion Criteria:

* Comorbidities, including type 1 diabetes, cardiovascular disease, thyroid disease, liver disease, kidney disease, cancer, mental disorders, and the use of drugs related to the aforementioned diseases,
* Pregnancy,
* Patients with a BMI over 35 who were on a weight loss diet or had taken weight loss supplements for less than 6 months
* A history of allergy to one of the components of the nestling fruit, carob leaf, carob fruit, alfalfa seed, fenugreek seed, lemon, Nettles and sumac and also
* Lactating women
* Regularly consuming cigarettes or alcohol
* Using psychiatric drugs or insulin
* Changing in the medication regimen during the trial period. For example, to start receiving insulin therapy, become pregnant, or no longer follow medication and dietary instructions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | Day 0, 15, 90, 180 post intervention
  Change in fasting blood glucose in response to intervention

SECONDARY OUTCOMES:
Insulin level | Day 0, 15, 90, 180 post intervention
  Change in insulin level in response to intervention
Hemoglobin A1c level | Day 0, 15, 90, 180 post intervention
  Change in hemoglobin A1c level in response to intervention
High density lipoprotein (HDL) level | Day 0, 15, 90, 180 post intervention
  Change in high density lipoprotein (HDL) level in response to intervention
Low density lipoprotein (LDL) level | Day 0, 15, 90, 180 post intervention
  Change in low density lipoprotein (LDL) level in response to intervention
Triglyceride level | Day 0, 15, 90, 180 post intervention
  Change in triglyceride level in response to intervention
Total cholesterol level | Day 0, 15, 90, 180 post intervention
  Change in total cholesterol level in response to intervention
Aspartate transaminase level | Day 0, 15, 90, 180 post intervention
  Change in aspartate transaminase level in response to intervention
Alanine aminotransferase level | Day 0, 15, 90, 180 post intervention
  Change in alanine aminotransferase level in response to intervention
Blood urea nitrogen level | Day 0, 15, 90, 180 post intervention
  Change in blood urea nitrogen level in response to intervention
Creatinine level | Day 0, 15, 90, 180 post intervention
  Change in creatinine level in response to intervention
Prothrombin time | Day 0, 15, 90, 180 post intervention
  Change in prothrombin time in response to intervention
Bilirubin level | Day 0, 15, 90, 180 post intervention
  Change in bilirubin level in response to intervention
Ferritin level | Day 0, 15, 90, 180 post intervention
  Change in ferritin level in response to intervention
Cholinesterase level | Day 0, 15, 90, 180 post intervention
  Change in cholinesterase level in response to intervention
High-sensitivity C-reactive protein level | Day 0, 15, 90, 180 post intervention
  Change in high-sensitivity C-reactive protein level in response to intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Reza hospital and clinic of Salamat, Tabriz, AzarbayejaneShargi, Iran